CLINICAL TRIAL: NCT04245579
Title: Cognitive Training in Elders Without Dementia Using UMAM Method. Genetic, Brain Volume and Cognitive Reserve Predictors: A Randomized Controlled Study
Brief Title: Effectiveness of a Cognitive Training Program (UMAM Method) in Elderly People Without Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madrid Salud (Other)
Collaborators: Universidad Complutense de Madrid (Other); Hospital San Carlos, Madrid (Other); Centro de Tecnología Biomédica, Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15/382-E_BS
Record Dates: First submitted 2019-12-22; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Age-Related Memory Disorders
Keywords: cognitive training; memory failures; APOE; brain volume; cognitive reserve
MeSH Terms: conditions — Memory Disorders

ARMS (2):
- Experimental Group (Experimental): The experimental group carried out a 30-session multi-factorial group memory training program (UMAM method), with a frequency of three weekly sessions of 90 minutes each. The training program consists of four modules: 1- Stimulation of cognitive processes; learning and practicing internal memory strategies and solving everyday forgetfulness; 2- Instruction in basic concepts about memory; 3- Intervention on daily living and forgetting experiences, using internal and external strategies to solve everyday memory failures; 4- Metacognition or metamemory: the subjects were to reflect about their cognitive failures by analyzing the causes and variables of those failures.
  In addition, the experimental group followed the standard activities in which all users attending the Center are involved (planned interviews, dialogue-conferences, general health recommendations, etc.).
  Interventions: Other: Multifactorial Memory Training Program (UMAM method)
- Control Group (No Intervention): The Control Group followed the standard activities in which all users attending the Center are involved (planned interviews, dialogue-conferences, general health recommendations, etc.).

INTERVENTIONS:
Other: Multifactorial Memory Training Program (UMAM method)
  Arms: Experimental Group

SUMMARY:
The study is oriented to analyze the effectiveness of a cognitive training method (UMAM) on cognitive functions, subjective memory and mood state in elderly people without dementia. On the other hand, the study aims to examine whether variables such as cognitive reserve (e.g. educational level), APOE genotype and intracranial volume are related to increased benefit after the intervention. The researchers hope to find that greater cognitive reserve, not having the APOE allele ε4, and a greater volume of memory-related brain areas, are associated with better outcomes after the cognitive intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years old.
* Having a global cognitive performance > 23 in the Mini Mental State Examination Test.
* Having no history of neurological or serious psychiatric disorders (severe psycho-affective disorders and psychosis or other psychiatric disorders like alcoholism).

Exclusion Criteria:

* Chronic use of anxiolytics.
* Chronic use of neuroleptics.
* Chronic use of anticonvulsants.
* Having hearing or vision impairments that would preclude testing.
* Magnetic Resonance Imaging (MRI) contraindications.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in general cognition | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in general cognition, assessed with the Mini Mental State Examination Test (MMSE) and the 7 Minutes Test (7M).The score ranges from 0 to 30 points (MMSE) and from 0 to 89 points (7M). In both cases, the higher scores indicate a better outcome.
Change in verbal memory | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in verbal memory, assessed with the Word List Test of the Wechsler Memory Scale-III. The score ranges from 0 to 48 points. Higher scores indicate a better outcome.
Change in logical memory | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in immediate and delayed logical memory, assessed with the Logical Memory Test (immediate and delayed units) of the Wechsler Memory Scale-III. The score ranges from 0 to 75 points (immediate units) and from 0 to 50 (delayed units). Higher scores indicate a better outcome.
Change in visual memory | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in visual memory, assessed with the Rey memory test (form B). The score ranges from 0 to 22 points. Higher scores indicate a better outcome.
Change in daily memory | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in daily memory, assessed with the Rivermead Behavioral Memory Test. The score ranges from 0 to 24 points. Higher scores indicate a better outcome.
Change in attentional amplitude | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in attentional amplitude, assessed with the Direct Digit Test of the Wechsler Memory Scale-III. The score ranges from 0 to 16 points. Higher scores indicate a better outcome.
Change in attentional control | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in attentional control, assessed with the Inverse Digit Test of the Wechsler Memory Scale-III. The score ranges from 0 to 14 points. Higher scores indicate a better outcome.
Change in attention and processing speed | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in attention, assessed with the Trail Making Test, form A. The score ranges from 0 to 200 points. Higher scores indicate a worse outcome.
Change in alternating attention and planning | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in alternating attention and planning, assessed with the Trail Making Test, form B. The score ranges from 0 to 400 points. Higher scores indicate a worse outcome.
Change in naming ability (language) | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in naming ability, assessed with the Boston Naming Test. The score ranges from 0 to 60 points. Higher scores indicate a better outcome.
Change in verbal fluency (language) | This cognitive variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in phonologic and semantic verbal fluency, assessed with the Phonological Verbal Fluency Test and the Semantic Fluency Test respectively. The score goes from zero onwards (there is no upper limit). Higher scores indicate a better outcome.
Change in subjective memory | This variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in Subjective Memory, assessed with the Memory Failures of Everyday Questionnaire.The score ranges from 0 to 56 points. Higher scores indicate a worse outcome.
Change in mood | This variable was assessed before and after the intervention. The interval between the pre and post-intervention assessment was 6 months.
  The measure of the post-intervention change in mood, assessed with the Geriatric Depression Scale. The score ranges from 0 to 15 points. Higher scores indicate a worse outcome.
The Cognitive Reserve as a predictor of change. | Cognitive Reserve was assessed in the pre-intervention assessment.
  The Cognitive Reserve was assessed with Rami Test. The score ranges from 0 to 25 points.
The Genetic Profile as a predictor of change. | The Genetic Profile was assessed in the pre-intervention assessment.
  The Genetic Profile was obtained by genetic analysis employing a blood test. APOE gene has been coded as 1 (meaning no ε4 allele), or 0 (for at least one ε4 allele).
The Brain Volume as a predictor of change. | The Brain Volume was assessed in the pre-intervention assessment.
  The Brain Volume (total gray volume, left hippocampus, right hippocampus and total intracranial volume) was assessed by magnetic resonance imaging. Unit of measure: mm3.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Prevención del Deterioro Cognitivo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montejo Carrasco P, Montenegro-Pena M, Prada Crespo D, Rodriguez Rojo I, Barabash Bustelo A, Montejo Rubio B, Marcos Dolado A, Maestu Unturbe F, Delgado Losada ML. APOE genotype, hippocampal volume, and cognitive reserve predict improvement by cognitive training in older adults without dementia: a randomized controlled trial. Cogn Process. 2024 Nov;25(4):673-689. doi: 10.1007/s10339-024-01202-3. Epub 2024 Jun 19. PMID 38896211